CLINICAL TRIAL: NCT01243697
Title: Assessment of Desogestrel for a Pharmacological Recovery of Ventilatory Activity in Congenital Central Hypoventilation Syndrome - Ondine Syndrome
Brief Title: Assessment of Desogestrel in Ondine Syndrome
Acronym: RESPIRONDINE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P101001
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2012-10

CONDITIONS: Ondine Syndrome
Keywords: Desogestrel; Chemosensitivity
MeSH Terms: conditions — Sleep Apnea, Central | interventions — Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- desogestrel (Experimental): Tablets of 75 µg, once daily during 112 days
  Interventions: Drug: desogestrel

INTERVENTIONS:
Drug: desogestrel — Tablets of 75 µg, once daily during 112 days

SUMMARY:
The congenital central hypoventilation syndrome (CCHS), also known as the Ondine syndrome, is a very rare genetic disorder. In contrast with healthy people, patients do not increase breathing in response to an excess of carbon dioxide (CO2). As a consequence, they do not breath sufficiently, or even stop breathing, during sleep. Their survival depends only on mechanical respiratory assistance, all life long.

We have recently published two cases of recovery of a response to CO2 in patients taking desogestrel as a contraceptive pill. The goal of the study is therefore to assess the hypothesis that desogestrel will restore a respiratory response to CO2 in CCHS patients and allow them to breath sufficiently during sleep without mechanical assistance.

DETAILED DESCRIPTION:
Rationale of the study The congenital central hypoventilation syndrome (CCHS), also called Ondine syndrome or Ondine's curse, is a rare orphan disease associated with mutations of the PHOX 2B gene. It is characterized by an absence or a deep reduction in the ventilatory response to hypercapnia and hypoxia. As a consequence, life-threatening hypoventilation or apneas occur during sleep and, in some patients, also during wakefulness. Survival thus depends on mechanical ventilatory assistance (or on phrenic pacing), all life long. There is no pharmacological treatment.

We have fortuitously observed two cases of recovery of ventilatory response to hypercapnia in patients taking desogestrel, a very potent progestin, as a contraceptive treatment ("Straus, C., et al. Respir. Physiol. Neurobiol. 2010 ; 171 : 171-174").

The hypothesis of the research project stems from these observations. It assumes that desogestrel will restore a chemosensitivity to hypercapnia in Ondine patients that will allow them to breath sufficiently without mechanical ventilatory assistance during sleep.

The primary goal of the study will be to assess whether a treatment with desogestrel will restore a ventilatory response to hypercapnia. The secondary goal will be to evaluate whether this response will allow the patients to be weaned from mechanical ventilatory assistance during sleep.

Methods The study will take place in one unique hospital, the Pitie-Salpetriere Hospital in Paris, France. It will be conducted in volunteer pubescent female patients. Patients with contra-indications to desogestrel will not be included.

The ventilatory response to hypercapnia will be assessed through the rebreathing method and through a blinded procedure specifically designed for the study. Sleep and breathing during sleep will be assessed through polysomnography. Blood gas analysis as well as hormonal and ionic analysis of the blood will be performed. The ventilatory response to hypoxia will also be assessed. Changes in cerebral activation will be looked for using functional magnetic resonance imaging (fMRI).

Protocol Patients will be first assessed with all the tests mentioned in the above paragraph, except fMRI. Polysomnography will be performed under mechanical ventilation.

Patients who will not take any contraceptive oral treatment with estrogens or progestin and whose response to hypercapnia will be low enough will immediately continue the study. An fMRI will be performed and the patients will be prescribed desogestrel 75 µg daily.

Patients who will be under an oral contraceptive treatment with estrogens or progestin will have to stop it and to use mechanical contraception (condom). All the patients taking an oral contraceptive treatment will be assessed after having stopped these drugs, with all the tests mentioned in the "methods" paragraph, except fMRI. Polysomnography will be performed under mechanical ventilation. If their ventilatory response to hypercapnia will be low enough an fMRI will be performed and the patients will be prescribed desogestrel 75 µg daily.

All the patients will be assessed under treatment with desogestrel. If the slope of the ventilatory response to hypercapnia is more than 1L/min/mmHg, an attempt of weaning from mechanical ventilation during sleep will replace the usual polysomnography under mechanical ventilation. The patients will be admitted in an intensive care unit where they will sleep without ventilatory assistance. Polysomnographic recordings will be performed with a portable device. In case of prolonged hypopneas or apneas or in case of arterial desaturation, patients will be awakened and mechanical ventilation will be resumed. The attempt of weaning will be regarded as a failure. In the absence of those criteria, the weaning will be regarded as a possible success. However, the investigators will not prescribe to the patient to sleep without ventilatory assistance. Their attending physician will have to take the final decision regarding this issue.

ELIGIBILITY:
Inclusion criteria :

* Ondine syndrome
* Pubescent female

Exclusion criteria :

* Contra-indications to a treatment with desogestrel.
* Other treatment with estrogens or progestin that cannot be stopped.

Ages: 10 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Increase in the ventilatory response to hypercapnia | 112 days

SECONDARY OUTCOMES:
Ventilatory response to hypoxia | 112 days
Activation of new cerebral regions in fMRI | 112 days
Weaning from mechanical ventilation during sleep | 112 days

CONTACTS AND LOCATIONS:
Overall Officials: STRAUS Christian, MD, PhD, Principal Investigator — Pitie Salpetriere Hospital (APHP)
Locations (1):
- Pitie salpetriere hospital, Paris, France

REFERENCES:
- [Derived] Sevoz-Couche C, Patout M, Charbit B, Similowski T, Straus C. Higher baseline heart rate variability in CCHS patients with progestin-associated recovery of hypercapnic ventilatory response. Respir Res. 2024 Feb 9;25(1):87. doi: 10.1186/s12931-023-02625-w. PMID 38336689
- [Derived] Sharman M, Gallea C, Lehongre K, Galanaud D, Nicolas N, Similowski T, Cohen L, Straus C, Naccache L. The cerebral cost of breathing: an FMRI case-study in congenital central hypoventilation syndrome. PLoS One. 2014 Sep 30;9(9):e107850. doi: 10.1371/journal.pone.0107850. eCollection 2014. PMID 25268234
- [Derived] Straus C, Similowski T. Congenital central hypoventilation syndrome and desogestrel: a call for caution: addendum to "C. Straus, H. Trang, M.H. Becquemin, P. Touraine, T. Similowski, Chemosensitivity recovery in Ondine's curse syndrome under treatment with desogestrel" [Respir. Physiol. Neurobiol. 171 (2010) 171-174]. Respir Physiol Neurobiol. 2011 Sep 15;178(2):357-8. doi: 10.1016/j.resp.2011.07.007. Epub 2011 Jul 23. PMID 21801857